CLINICAL TRIAL: NCT03817697
Title: Analysis of Non-vaccination Factors Against Hepatitis B Virus (HBV) in Drug Users Consulting at the Croix-rousse Drug Addict Care Center (Annuaire Centres de Soins, d'Accompagnement et de prévention en Addictologie (CSAPA))
Brief Title: Non-vaccination Factors Against Hepatitis B Virus in Drug Users
Acronym: ANOVAC B
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL18_0992; 2019-A00114-53 (Other: ID-RCB)
Record Dates: First submitted 2019-01-23; First posted 2019-01-25 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Adult Patients Drug Users; Substituted / Weaned or Not
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Drug users: The cohort will be constituted of adult patients drug users, substituted/weaned or not, consulting at the Croix-Rousse CSAPA
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — The socio-demographic characteristics of patients, their current and past drug use as well as their knowledge of hepatitis B and vaccination, will be collected via a questionnaire, conducted by the service's addictologists at the beginning of the consultation.

SUMMARY:
Hepatitis B is one of the major public health problems in the world. According to World Health Organization (WHO) data, about 2 billion people have been in contact with the hepatitis B virus (HBV), and 257 million have chronic HBV infection.

Although France is a low endemic country, with just over 280,000 people with chronic infection, hepatitis B remains a public health problem due to its morbidity and mortality.

Drug users are a population at risk by their consumption practices (injection or sniffing), but also by other high-risk behaviours, particularly sexual behaviours.

Prevention therefore involves securing consumption practices (sterile and single-use equipment) and protection of sexual intercourse, but also by vaccination (protecting more than 90%).

Since 1982, HAS has recommended to systematically vaccinate drug users. However, according to the Marmottan study published in 2003, immunization coverage among drug addicts was already insufficient in 1999 (45.3%) and decreased again in 2000 and 2001 (15.6 and 21.7%).

This decrease can be explained by the controversy around the potential link, now refuted, between vaccine against HBV and demyelination, which has stopped the mass vaccination campaign launched by the French health authorities in 1995.

A study conducted between 2009 and 2012 on injecting drug users in Alsace, estimated vaccination coverage at 28%.

The hypothesize is that despite the recommendations in a population at high risk of contamination, and a balance of benefits and risks in favor of vaccination, vaccination coverage against the hepatitis B virus remains insufficient among drug users because of poor vaccination acquaintance, and hepatitis B in general, in this population.

Principal objective of this study is to identify non-vaccination factors against hepatitis B virus among drug users consulting at the Croix-Rousse CSAPA.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age ≥ 18 years)
* Patients with an addiction with product, substituted / weaned or not
* Patients consulting at the CSAPA of the Croix-Rousse hospital

Exclusion Criteria:

* Patients with an addiction without a product
* Patients who have never snorted or injected psychoactive product
* Patients protected by the law
* Patient refusing to participate to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients drug users, substituted / weaned or not, consulting at the Croix-Rousse CSAPA
Sampling Method: Non-Probability Sample
Enrollment: 137 (Actual)
Dates: Start 2019-04-10 (Actual); Primary Completion 2019-09-04 (Actual); Study Completion 2019-09-04 (Actual)

PRIMARY OUTCOMES:
comparison of the characteristics of patients vaccinated and unvaccinated against hepatitis B | One day
  These data will be collected via a questionnaire with questions of patient socio-demographic characteristics, as well as their knowledge of hepatitis B and vaccination.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital de la Croix-Rousse, 103 grande rue de la Croix-Rousse, Lyon, France

IPD SHARING:
Plan to Share IPD: No